CLINICAL TRIAL: NCT05495204
Title: External Comparison of Effectiveness of Ibalizumab in Clinical Trials vs. Other HTE Regimens in OPERA
Brief Title: External Comparison of Ibalizumab in Trials vs. Other Regimens in OPERA
Status: Completed | Type: Observational
Sponsor: Epividian (Industry)
Collaborators: Theratechnologies (Industry); FIECON (Unknown)
Responsible Party: Sponsor
Other Study IDs: COL2022-001
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: HIV-1-infection
Keywords: Heavily treatment experienced; External comparison; Ibalizumab; Virologic effectiveness
MeSH Terms: interventions — ibalizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBA+OBR (trials): Participants in TMB-202 or TMB-301/311 trials who received 800 mg ibalizumab every 2 weeks, with or without a loading dose
  Interventions: Drug: Ibalizumab
- Non-IBA+OBR (OPERA): Heavily treatment experienced adults living with HIV in care in OPERA, with documented resistance to ≥1 ARV from each of three ARV classes switching to a new regimen that does not include ibalizumab

INTERVENTIONS:
Drug: Ibalizumab — Participation in clinical trials vs. routine care in OPERA
  Other Names: Regimens not containing ibalizumab
  Groups: IBA+OBR (trials)

SUMMARY:
Among heavily treatment experienced people living with HIV, the virologic effectiveness of ibalizumab + optimized background regimen from two clinical trials will be compared to non-ibalizumab-containing regimens in routine clinical care in the OPERA cohort.

DETAILED DESCRIPTION:
The US Department of Health and Human Services (DHHS) HIV treatment guideline suggest that ibalizumab may be considered in the context of multidrug resistance without fully active ART options. However, clinical trials assessing ibalizumab efficacy did not include an active comparison arm in which participants did not receive ibalizumab. The use of external controls can provide valuable information and context to interpret the results of clinical trials when randomization to a control arm cannot be performed.

The OPERA (Observational Pharmaco-Epidemiology Research & Analysis) cohort, a large US electronic health record database, is well suited for this as the OPERA and trials populations arose from the same geographic location (i.e., US). An external comparison of ibalizumab + optimized background regimen from trials vs. non-ibalizumab containing regimens in routine clinical care in the OPERA cohort may confirm results from prior studies suggesting viral control benefits of ibalizumab.

ELIGIBILITY:
Inclusion Criteria (Trial IBA+OBR group):

* Participant in TMB-202 or TMB-301/311
* Received 800 mg IBA every 2 weeks, with or without a loading dose

Inclusion Criteria (OPERA non-IBA OBR group):

* HIV-1 infection
* 18 years or older
* Heavily treatment experienced (i.e., ever on a regimen containing either DTG BID or DRV BID)
* Documented resistance to ≥1 ARV from each of three ARV classes
* Genotype information available for all the relevant gene regions (see Table 2)
* Viral load > 200 copies/mL at index regimen initiation
* Not pregnant at index
* No new AIDS defining event within 3 months before/on index (except cutaneous Kaposi's sarcoma or HIVAW)
* No new cancer diagnosis within 12 weeks before/on index
* No IBA prescribed prior to/with the index regimen
* Index regimen does not include cabotegravir, fostemsavir, investigational drugs
* Viral sensitivity/susceptibility to at least one ARV in the index regimen
* Baseline VL available (within 6 months before/at index)
* Baseline CD4 available (within 6 months before/at index)
* ≥1 VL measurement at any time after index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All TMB-202 and TMB-301/311 trial participants randomized to 800 mg IBA every 2 weeks with or without a loading dose will be included in the main analyses. From the OPERA cohort, adult PWH with resistance from three ARV classes will be considered for inclusion. People with HIV in OPERA initiating a new non-IBA OBR between 01JAN2008 and 31DEC2020 will be included; person-time will be censored at the first of (a) initiation of a select potent ARV, (b) >45 days without ART, (c) 12 months after last clinical contact, (d) death, or (e) study end.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Viral suppression | Week 24
  Viral load <200 copies/mL
Viral suppression | Week 48
  Viral load <200 copies/mL
Viral suppression | Week 60
  Viral load <200 copies/mL
Viral suppression | Week 96
  Viral load <200 copies/mL
Viral undetectability | Week 24
  Viral load <50 copies/mL
Viral undetectability | Week 48
  Viral load <50 copies/mL
Viral undetectability | Week 60
  Viral load <50 copies/mL
Viral undetectability | Week 96
  Viral load <50 copies/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Epividian, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT05495204/Prot_SAP_000.pdf